CLINICAL TRIAL: NCT03144700
Title: The Natural History and Prognostic Factors of Compensated Cirrhosis: An Ambi Prospective Cohort Study
Brief Title: The Natural History and Prognostic Factors of Compensated Cirrhosis.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Cirrhosis-11
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Compensated Cirrhosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Compensated Cirrhosis

SUMMARY:
Study Design and Methodology

* Study Population:Compensated Cirrhosis
* Study Design: An Ambi Prospective Cohort study
* Study Period: 2 Years
* Sample size: Retrospective- All patients from Jan 2010 to Mar 2017 Prospective- Assuming the incidence of clinical decompensation is 5%/year.With alpha of 5%, power 80% we need to enroll 138 cases. Further assuming 20% drop out 166 cases will be enrolled.
* Intervention: This is an observational study. No intervention will be given.

Monitoring and assessment: All the routine investigation and clinical information will be collected at 6, 12,18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years
2. Compensated cirrhosis
3. Biopsy proven cirrhosis or LSM > 12.5 Kpa.

Exclusion Criteria:

1. Any current or prior clinical decompesnation (ascites, jaundice, encephalopathy or gastrointestinal hemorrhage).
2. Pregnant Women
3. Hepatocellular Carcinoma
4. Known case of severe cardiopulmonary disease
5. Known case of severe Hepato Pulmonary Syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Compensated Cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Development of ascites, jaundice, encephalopathy or gastrointestinal hemorrhage) during the follow up period of 2 yeas | 2 years

SECONDARY OUTCOMES:
Patients with new onset/progression of esophageal varices during the period of 2 years | 2 years
Reduction in portal pressure with >20% from baseline at 6 months | 6 months
Reduction in portal pressure with >20% from baseline at 1 year | 1 year
Reduction in portal pressure with >20% from baseline at 2 year. | 2 year
Survival during the period of 2 years. | 2 years
Number of patients develop hepatocellular carcinoma (HCC) during follow up period 2 years. | 2 years
Number of patients develop Pulmonary Syndrome (HPS) during follow up period of 2 years. | 2 years
Number of patients develop Minimal Hepatic Encephalopathy (MHE) during follow up period of 2 years. | 2 years
Number of patients develop Hypersplenism during follow up period of 2 years. | 2 years
Number of patients develop Hepatic osteodystrophy during follow up period of 2 years. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No